CLINICAL TRIAL: NCT00575133
Title: Multicentric, Prospective, Non-interventional, Long-term Cohort Study in Patients With Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Prospective Cohort Study in Patients With NAFLD
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EK-1450
Record Dates: First submitted 2007-11-26; First posted 2007-12-18 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsy
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the importance of intracellular signalling pathways and its deregulation in adiposity and diabetes-related insulin resistance, liver tissue samples of patients suffering from non-alcoholic fatty liver disease (NAFLD) and non-alcoholic steatohepatitis (NASH)will be analyzed prospectively from a liver tissue bank.

DETAILED DESCRIPTION:
Patients with suspected fatty liver disease will be screened (and excluded in the presence) of alternative clinical condition associated with NAFLD (see exclusion criteria). Of all patients fulfilling inclusion criteria, relevant baseline characteristics (incl. epidemiological, physiological and biochemical data) will be obtained. In addition, radiological examination will be performed using sonography and fibroscan to assess non-invasively the individual extent of hepatic fat deposition, liver stiffness (fibrosis) and amount of visceral fat mass. In case of high clinical, laboratory and radiological suspicion for NAFLD, a diagnostic liver biopsy will be performed. A part of the liver tissue is used for histological confirmation of NAFLD and subsequent grading and staging according established criteria. Parts of the remaining liver tissue will be stored for later molecular and histological analysis. In addition, several serum samples are collected of patients and stored for future analysis. All patients will be followed up annually (incl. physical examination, metabolic characterisation, clinical chemistry and liver sonography) and additional serum samples will be collected for future analysis. Liver biopsy is not repeated after defined time period, but in case of clinical evidence for disease progression.

ELIGIBILITY:
Inclusion criteria:

* Patients with histologically confirmed fatty liver disease

Exclusion criteria:

* History of significant alcohol consumption
* Viral hepatitis
* Autoimmune hepatitis
* Metabolic diseases (e.g. hemochromatosis, M. Wilson, alpha 1-antitrypsin deficiency)
* Hepatotoxic medication (e.g. amiodarone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-alcoholic fatty liver disease
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2007-12; Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Disease regression/progression | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Giatgen Spinas, Prof. MD, Principal Investigator — University Hospital Zurich, Endocrinology and Diabetology
Locations (1):
- University Hospital Zurich, Endocrinology and Diabetology, Zurich, Canton of Zurich, Switzerland